CLINICAL TRIAL: NCT01827462
Title: Immune Senescence in the Elderly: Comparison of Immune Responses to Influenza Vaccine In Adults of Different Ages
Brief Title: Comparison of Immune Responses to Influenza Vaccine In Adults of Different Ages (SLVP015 2007-2017)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Cornelia L. Dekker, Professor, Pediatrics, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SU-03192011-7599; 1U19AI090019-01 (NIH); 51731 (Other: Bill and Melinda Gates Foundation); AG-NS-0792-11 (Other: Ellison Foundation)
Record Dates: First submitted 2013-04-04; First posted 2013-04-09 (Estimated); Results first posted 2017-06-12 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Influenza
Keywords: Inactivated, trivalent influenza vaccine; elderly; immunosenescence; longitudinal study; Inactivated, High-Dose trivalent influenza vaccine; Inactivated, quadrivalent influenza vaccine; young adults
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 18-30 year olds at enrollment (Experimental): Licensed seasonal Fluzone (inactivated influenza vaccine):
  Trivalent, inactivated influenza vaccine (TIV) was given through the 2013-2014 season.
  Beginning with 2014-2015 season, Quadrivalent, inactivated influenza vaccine (IIV4) was given.
  Interventions: Biological: Trivalent, inactivated influenza vaccine (TIV); Biological: Quadrivalent, inactivated influenza vaccine (IIV4)
- 60-80 year olds at enrollment (Experimental): Licensed seasonal Fluzone (inactivated influenza vaccine):
  Trivalent, inactivated influenza vaccine (TIV) was given through the 2013-2014 season.
  Beginning with 2014-2015 season, High-Dose trivalent, inactivated influenza vaccine (TIV High-Dose) was given.
  Interventions: Biological: Trivalent, inactivated influenza vaccine (TIV); Biological: High-Dose Trivalent, inactivated influenza vaccine (TIV High-Dose)
- 80-100 year olds at enrollment (Experimental): Licensed seasonal Fluzone (inactivated influenza vaccine):
  Trivalent, inactivated influenza vaccine (TIV) was given through the 2013-2014 season.
  Beginning with 2014-2015 season, High-Dose trivalent, inactivated influenza vaccine (TIV High-Dose) was given.
  Interventions: Biological: Trivalent, inactivated influenza vaccine (TIV); Biological: High-Dose Trivalent, inactivated influenza vaccine (TIV High-Dose)

INTERVENTIONS:
Biological: Trivalent, inactivated influenza vaccine (TIV) — Licensed Seasonal Influenza Vaccine TIV
  Other Names: Fluzone (IM)
Biological: Quadrivalent, inactivated influenza vaccine (IIV4) — Licensed Seasonal Influenza Vaccine IIV4
  Other Names: Fluzone (IM)
  Arms: 18-30 year olds at enrollment
Biological: High-Dose Trivalent, inactivated influenza vaccine (TIV High-Dose) — Licensed Seasonal High-Dose Influenza Vaccine TIV
  Other Names: Fluzone High-Dose (IM)
  Arms: 60-80 year olds at enrollment; 80-100 year olds at enrollment

SUMMARY:
In this study the investigators are trying to understand how immune function declines in the elderly using annual influenza vaccinations as a model system. The longitudinal study began in 2007 and continued through early 2017.

DETAILED DESCRIPTION:
Participants ranging in age from 18 to 100 at time of initial enrollment will be immunized annually with the seasonal influenza vaccine, Fluzone, on Day 0. Follow-up visits will be conducted on Day 6-8 and Day 28. Unsolicited adverse events are collected from immunization until the Day 28 visit, serious adverse events are collected for the entire time of study participation. A blood sample is collected pre-immunization and at each follow-up visit. Volunteers will be followed for up to 11 years, those too frail to come in for visits received annual phone calls to monitor health. Last annual influenza vaccines were given in Fall 2015.

The main basic research effort will be to collect safety data and follow medical history events in elderly and younger control subjects. Investigators will also look at immune responses to influenza vaccination. In 2008, 2012 and 2014, the cohort added additional participants to replace those who had withdrawn.

Beginning in 2014, those participants 65 years and older were immunized with High Dose trivalent Fluzone and younger participants received the quadrivalent formulation of Fluzone.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-30, 60-79, or 80-100 years, inclusive at time of initial enrollment
* General good health and ambulatory at time of enrollment
* No acute illness at time of vaccination
* Willing and able to sign Informed Consent
* Available for follow-up for the planned duration of the study
* Acceptable medical history by screening evaluation and brief clinical assessment
* All female subjects of childbearing potential must use an acceptable method of contraception and not become pregnant for the duration of the clinical phase of the study (approximately 1 month to completion of Visit 3). (Acceptable contraception may include implants, injectables, combined oral contraceptives, effective intrauterine devices (IUDs), sexual abstinence, or a vasectomized partner).

Exclusion Criteria:

* Prior off-study vaccination with trivalent or quadrivalent (depending no year) influenza vaccine (TIV or IIV4) or live attenuated influenza vaccine (LAIV) in the current flu season
* Allergy to egg or egg products
* Allergy to vaccine components, including thimerosal
* Active systemic or serious concurrent illness, including febrile illness on the day of vaccination
* History of immunodeficiency
* Any chronic disorder which, in the opinion of the investigator, might jeopardize volunteer safety or compliance with the protocol.
* Blood pressure >150 systolic or > 95 diastolic at Visit 1
* Chronic Hepatitis B or C.
* Recent or current use of systemic immunosuppressive medication, including glucocorticoids (corticosteroid nasal sprays and inhaled steroids are permissible). Use of oral steroids (<20mg prednisone-equivalent/day) may be acceptable after review by the investigator.
* Autoimmune disease (including rheumatoid arthritis treated with immunosuppressive medication such as Plaquenil, methotrexate, prednisone, Enbrel) which, in the opinion of the investigator, might jeopardize volunteer safety or compliance with the protocol.
* History of blood dyscrasias or hemoglobinopathies requiring regular medical follow up or hospitalization during the preceding year
* Use of anti-coagulation medication such as Coumadin or Lovenox, or anti-platelet agents such as aspirin, Plavix, Aggrenox must be reviewed by investigator to determine if this would affect the volunteer's safety.
* Receipt of blood or blood products within the past 6 months
* Medical or psychiatric condition or occupational responsibilities that preclude subject compliance with the protocol
* Receipt of inactivated vaccine within 14 days prior to vaccination
* Receipt of live, attenuated vaccine within 60 days of vaccination
* History of Guillain-Barré Syndrome
* Pregnant or lactating woman
* Use of investigational agents within 30 days prior to enrollment
* Donation of the equivalent of a unit of blood within 6 weeks prior to enrollment
* Any condition which, in the opinion of the investigator, might interfere with volunteer safety, study objectives or the ability of the participant to understand or comply with the study protocol.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2007-10 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia L Dekker, MD, Principal Investigator — Stanford University; Mark M Davis, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The NIH Human Immunology Project Consortium (HIPC) data repositories (ImmPORT) may store the results of the research assays results. Genetic data that is developed in this study may be made available to other researchers through the National Center for Biotechnology Information (NCBI) databases. Results from research assays will be labeled with a unique ID code and the volunteer identity (except for age) will not be disclosed.

REFERENCES:
- [Background] Furman D, Jojic V, Kidd B, Shen-Orr S, Price J, Jarrell J, Tse T, Huang H, Lund P, Maecker HT, Utz PJ, Dekker CL, Koller D, Davis MM. Apoptosis and other immune biomarkers predict influenza vaccine responsiveness. Mol Syst Biol. 2013 Apr 16;9:659. doi: 10.1038/msb.2013.15. PMID 23591775
- [Background] Price JV, Jarrell JA, Furman D, Kattah NH, Newell E, Dekker CL, Davis MM, Utz PJ. Characterization of influenza vaccine immunogenicity using influenza antigen microarrays. PLoS One. 2013 May 29;8(5):e64555. doi: 10.1371/journal.pone.0064555. Print 2013. PMID 23734205
- [Background] Wang C, Liu Y, Xu LT, Jackson KJ, Roskin KM, Pham TD, Laserson J, Marshall EL, Seo K, Lee JY, Furman D, Koller D, Dekker CL, Davis MM, Fire AZ, Boyd SD. Effects of aging, cytomegalovirus infection, and EBV infection on human B cell repertoires. J Immunol. 2014 Jan 15;192(2):603-11. doi: 10.4049/jimmunol.1301384. Epub 2013 Dec 11. PMID 24337376
- [Background] Furman D, Hejblum BP, Simon N, Jojic V, Dekker CL, Thiebaut R, Tibshirani RJ, Davis MM. Systems analysis of sex differences reveals an immunosuppressive role for testosterone in the response to influenza vaccination. Proc Natl Acad Sci U S A. 2014 Jan 14;111(2):869-74. doi: 10.1073/pnas.1321060111. Epub 2013 Dec 23. PMID 24367114
- [Background] Jackson KJ, Liu Y, Roskin KM, Glanville J, Hoh RA, Seo K, Marshall EL, Gurley TC, Moody MA, Haynes BF, Walter EB, Liao HX, Albrecht RA, Garcia-Sastre A, Chaparro-Riggers J, Rajpal A, Pons J, Simen BB, Hanczaruk B, Dekker CL, Laserson J, Koller D, Davis MM, Fire AZ, Boyd SD. Human responses to influenza vaccination show seroconversion signatures and convergent antibody rearrangements. Cell Host Microbe. 2014 Jul 9;16(1):105-14. doi: 10.1016/j.chom.2014.05.013. Epub 2014 Jun 26. PMID 24981332
- [Background] Furman D, Jojic V, Sharma S, Shen-Orr SS, Angel CJ, Onengut-Gumuscu S, Kidd BA, Maecker HT, Concannon P, Dekker CL, Thomas PG, Davis MM. Cytomegalovirus infection enhances the immune response to influenza. Sci Transl Med. 2015 Apr 1;7(281):281ra43. doi: 10.1126/scitranslmed.aaa2293. PMID 25834109
- [Background] Looney TJ, Lee JY, Roskin KM, Hoh RA, King J, Glanville J, Liu Y, Pham TD, Dekker CL, Davis MM, Boyd SD. Human B-cell isotype switching origins of IgE. J Allergy Clin Immunol. 2016 Feb;137(2):579-586.e7. doi: 10.1016/j.jaci.2015.07.014. Epub 2015 Aug 22. PMID 26309181
- [Background] Haddon DJ, Jarrell JA, Diep VK, Wand HE, Price JV, Tangsombatvisit S, Credo GM, Mackey S, Dekker CL, Baechler EC, Liu CL, Varma M, Utz PJ. Mapping epitopes of U1-70K autoantibodies at single-amino acid resolution. Autoimmunity. 2015;48(8):513-23. doi: 10.3109/08916934.2015.1077233. Epub 2015 Aug 31. PMID 26333287
- [Background] Shen-Orr SS, Furman D, Kidd BA, Hadad F, Lovelace P, Huang YW, Rosenberg-Hasson Y, Mackey S, Grisar FA, Pickman Y, Maecker HT, Chien YH, Dekker CL, Wu JC, Butte AJ, Davis MM. Defective Signaling in the JAK-STAT Pathway Tracks with Chronic Inflammation and Cardiovascular Risk in Aging Humans. Cell Syst. 2016 Oct 26;3(4):374-384.e4. doi: 10.1016/j.cels.2016.09.009. Epub 2016 Oct 13. PMID 27746093
- [Background] Furman D, Chang J, Lartigue L, Bolen CR, Haddad F, Gaudilliere B, Ganio EA, Fragiadakis GK, Spitzer MH, Douchet I, Daburon S, Moreau JF, Nolan GP, Blanco P, Dechanet-Merville J, Dekker CL, Jojic V, Kuo CJ, Davis MM, Faustin B. Expression of specific inflammasome gene modules stratifies older individuals into two extreme clinical and immunological states. Nat Med. 2017 Feb;23(2):174-184. doi: 10.1038/nm.4267. Epub 2017 Jan 16. PMID 28092664
- [Background] de Bourcy CF, Angel CJ, Vollmers C, Dekker CL, Davis MM, Quake SR. Phylogenetic analysis of the human antibody repertoire reveals quantitative signatures of immune senescence and aging. Proc Natl Acad Sci U S A. 2017 Jan 31;114(5):1105-1110. doi: 10.1073/pnas.1617959114. Epub 2017 Jan 17. PMID 28096374
- [Background] Kay AW, Bayless NL, Fukuyama J, Aziz N, Dekker CL, Mackey S, Swan GE, Davis MM, Blish CA. Pregnancy Does Not Attenuate the Antibody or Plasmablast Response to Inactivated Influenza Vaccine. J Infect Dis. 2015 Sep 15;212(6):861-70. doi: 10.1093/infdis/jiv138. Epub 2015 Mar 4. PMID 25740957
- [Background] Roskin KM, Simchoni N, Liu Y, Lee JY, Seo K, Hoh RA, Pham T, Park JH, Furman D, Dekker CL, Davis MM, James JA, Nadeau KC, Cunningham-Rundles C, Boyd SD. IgH sequences in common variable immune deficiency reveal altered B cell development and selection. Sci Transl Med. 2015 Aug 26;7(302):302ra135. doi: 10.1126/scitranslmed.aab1216. PMID 26311730
- [Background] Fang F, Yu M, Cavanagh MM, Hutter Saunders J, Qi Q, Ye Z, Le Saux S, Sultan W, Turgano E, Dekker CL, Tian L, Weyand CM, Goronzy JJ. Expression of CD39 on Activated T Cells Impairs their Survival in Older Individuals. Cell Rep. 2016 Feb 9;14(5):1218-1231. doi: 10.1016/j.celrep.2016.01.002. Epub 2016 Jan 28. PMID 26832412
- [Derived] Ju CH, Blum LK, Kongpachith S, Lingampalli N, Mao R, Brodin P, Dekker CL, Davis MM, Robinson WH. Plasmablast antibody repertoires in elderly influenza vaccine responders exhibit restricted diversity but increased breadth of binding across influenza strains. Clin Immunol. 2018 Aug;193:70-79. doi: 10.1016/j.clim.2018.01.011. Epub 2018 Feb 2. PMID 29410330
- See also: Stanford Institute for Immunity, Transplantation and Infection — http://iti.stanford.edu/

RESULTS

PARTICIPANT FLOW:
Groups:
- 18-30 Years Old at Enrollment; 60-79 Years Old at Enrollment; 80-100 Years Old at Enrollment: Participants receive the licensed annual trivalent vaccine, Fluzone®
  This vaccine is given intramuscularly
Period: Overall Study
Arm/Group | 18-30 Years Old at Enrollment | 60-79 Years Old at Enrollment | 80-100 Years Old at Enrollment
Started | 59 | 37 | 40
Completed | 18 | 19 | 12
Not Completed | 41 | 18 | 28

BASELINE CHARACTERISTICS:
Groups:
- 18-30 Years Old at Enrollment: Participants receive the licensed annual, Fluzone®
  This vaccine is given intramuscularly
- 60-79 Years Old at Enrollment: Participants receive the licensed annual vaccine, Fluzone®
  This vaccine is given intramuscularly
- 80-100 Years Old at Enrollment: Participants receive the licensed annual vaccine, Fluzone® or High Dose Fluzone®
  This vaccine is given intramuscularly
- Total: Total of all reporting groups
Arm/Group | 18-30 Years Old at Enrollment | 60-79 Years Old at Enrollment | 80-100 Years Old at Enrollment | Total
Number analyzed (Participants) | 59 | 37 | 40 | 136
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.6 (2.9) | 73.3 (5.0) | 89.5 (4.3) | 70.9 (23.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 22 | 26 | 78
  Male | 29 | 15 | 14 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 0 | 0 | 6
  Not Hispanic or Latino | 53 | 37 | 40 | 130
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 12 | 0 | 1 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 37 | 37 | 37 | 111
  More than one race | 8 | 0 | 2 | 10
  Unknown or Not Reported | 2 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 59 | 37 | 40 | 136

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Received the Influenza Vaccine
Time Frame: Day 0 annually while on study
Measure: Count of Participants; unit: Participants
Arm/Group | 18-30 Years Old at Enrollment | 60-79 Years Old at Enrollment | 80-100 Years Old at Enrollment
Number analyzed (Participants) | 59 | 37 | 40
Participants | 59 | 37 | 40

2. Secondary Outcome: Number of Participants With Related Adverse Events
Description: Related adverse events were recorded annually during this 10 year longitudinal study.
Time Frame: Day 0 to Day 28 following each annual vaccination while on study
Measure: Count of Participants; unit: Participants
Groups:
- 18-30 Years Old at Enrollment: Participants receive the licensed annual trivalent vaccine, Fluzone® through 2013-2014 then received licensed annual quadrivalent Fluzone.
  This vaccine is given intramuscularly
- 60-79 Years Old at Enrollment; 80-100 Years Old at Enrollment: Participants receive the licensed annual trivalent vaccine, Fluzone® through the 2013-2014 season. For the following seasons, they received Fluzone High-Dose.
  This vaccine is given intramuscularly
Arm/Group | 18-30 Years Old at Enrollment | 60-79 Years Old at Enrollment | 80-100 Years Old at Enrollment
Number analyzed (Participants) | 59 | 37 | 40
Participants
  Erythema at injection site | 0 | 0 | 1
  Rash at injection site | 0 | 0 | 1
  Pain at injection site | 1 | 0 | 0
  Flushing | 0 | 1 | 0
  High White Blood Cell Count | 0 | 1 | 0
  Lymphopenia | 0 | 0 | 1
  Thrombocytopenia | 1 | 0 | 0
  No Related Adverse Events | 57 | 35 | 37

3. Other Pre Specified Outcome: Evaluate Changes in Cytokine Profile in the Immune Response From Day 0 to Day 5-7 for T Cells and Antibody-secreting Cells (ASCs)
Time Frame: Day 0 to 7
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Evaluate Changes in Cytokine Profile in the Immune Response From Day 0 to Day 28-32 for Responses to the Vaccine Antigens
Time Frame: Day 0-Day28
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Unsolicited adverse events were reported during the 28 day period following each annual immunization. Serious adverse events were reported on an annual basis for this 10 year longitudinal study.
Description: Because serious adverse events were reported on an annual basis for this 10 year longitudinal study, individual participants often had multiple different adverse events over the course of their participation.
Groups:
- 18-30 Years Old at Enrollment: Participants receive the licensed annual trivalent vaccine, Fluzone® through the 2013-2014 season then they received licensed quadrivalent vaccine, Fluzone starting with the 2014-2015 season.
  This vaccine is given intramuscularly
- 60-79 Years Old at Enrollment; 80-100 Years Old at Enrollment: Participants receive the licensed annual trivalent vaccine, Fluzone® through the 2013-2014 season then they received licensed High-Dose trivalent inactivated vaccine, Fluzone High-Dose, starting with the 2014-2015 season.
  This vaccine is given intramuscularly
Arm/Group | 18-30 Years Old at Enrollment | 60-79 Years Old at Enrollment | 80-100 Years Old at Enrollment
All-Cause Mortality (participants affected / at risk) | 0/59 | 2/37 | 16/40
Serious Adverse Events (participants affected / at risk) | 2/59 | 20/37 | 34/40
Other Adverse Events (participants affected / at risk) | 31/59 | 29/37 | 21/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 18-30 Years Old at Enrollment (N=59) | 60-79 Years Old at Enrollment (N=37) | 80-100 Years Old at Enrollment (N=40)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3)
Congestive Heart Failure (Cardiac disorders) | 0 (0) | 1 (1) | 6 (6)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 2 (2) | 2 (2)
Hypetension (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Chest Pain (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Calcium Channel Blocker Overdose (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Syncopal Episode (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0)
Death (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3) — CHF
Ulcer (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea/Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diminished Cognition (General disorders) | 0 (0) | 1 (1) | 0 (0)
Weakness Worsening (General disorders) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1) — Family reported death due to old age
Death (General disorders) | 0 (0) | 0 (0) | 1 (1) — Family reported death due to advanced Alzheimer's
Death (General disorders) | 0 (0) | 0 (0) | 1 (1) — Cause not determined.
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Prosthetic Hip Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (3)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Systemic Inflammatory Response Syndrone (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Scabies (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Death (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) — Sepsis
Alcohol Detoxification (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Fractures/Accidents (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 3 (6) — Surgery was not required with these fractures. All fractures due to falls or car collisions.
Contusions/observation/hit by car (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Degenerative Joint Disease-pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Pancreatic Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) — Pancreatic Cancer
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) — Lung Canceer
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) — Ovarian Cancer
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) — Neuroendocrine Cancer
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) — GI malignancy
Parkinson's (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncopal Episode (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
UTI (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (3)
Urosepsis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 5 (7)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural Effusions/bilateral (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
COPD (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Appendectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 1 (1)
Hip Arthroplasty (Surgical and medical procedures) | 0 (0) | 2 (4) | 7 (9) — Due to osteoarthritis, revision for failed hip arthroplasty (3), Avascular Necrosis (1), fall (1)
Knee Arthroplasty (Surgical and medical procedures) | 0 (0) | 2 (3) | 0 (0) — Due to osteoarthritis -3
Bladder resection/transurethral (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) — Surgery performed for Bladder Cancer
Diaphragmatic Hernia Repair (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Microdiskectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) — Spinal stenosis
Pancreatoduodenectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) — Surgery performed for Ampulla Cancer
Perforated Pylric Ulcer repair (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) — Laparoscopic repair
Inguinal Hernia Repair (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1)
Pacemaker Placement (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1) — Due to Atrial Fibrillaiton
Node Ablation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) — Due to Atrial Tachycardia
Hemicolectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) — Laparoscopic repair of recurrent cecal polyp-right hemicolectomy with ileotranverse anastomosis
Aortic Valve Replacement (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Arthrectomy-Femoral Artery (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) — Claudication/PVD
Decompression of Lumbar Stenosis (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Femur Fracture Repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 2 (2) — Surgical repair of Intertronchanteric femur fracture due to fall (2).
Cardioversion (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) — Elective for Atrial Fibrillation
Cholecystectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) — Peformed for cholelithiasis
Colectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) — Surgery performed due to colon mass-Subtotal Colectomy with ileo-transverse colon anastomosis
Pancreatic Stent Placement (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1) — Obstruction due to pancreatic CA
Biliary Stent Placement (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1) — Obstruction due to pancreatic CA
Inferior Vena Cava Filter (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) — IVC filter placed as a precaution
Venoplasty (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) — Right subclavian and brachiocephalic veins due to RUE thrombus
Diverticulectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) — Zenker's diverticulum
Ankle Fracture (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) — Surgical repair of ankle fracture due to fall
Amnesia-Tansient (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Stroke (Vascular disorders) | 0 (0) | 2 (2) | 3 (3)
Subarachnoid Hemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) — Secondary to falls
Death (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) — Subdural Hematoma
Death (Vascular disorders) | 0 (0) | 1 (1) | 2 (2) — Stroke
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 18-30 Years Old at Enrollment (N=59) | 60-79 Years Old at Enrollment (N=37) | 80-100 Years Old at Enrollment (N=40)
Upper respiratory infection (Infections and infestations) | 14 (15) | 15 (17) | 5 (5)
Influenza Type Illness (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 2 (3) | 0 (0)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 1 (1) | 1 (1)
Lower Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 3 (3)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 4 (4)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 2 (3) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No